CLINICAL TRIAL: NCT01493960
Title: A Placebo-controlled, Double-blind, Randomised Study to Assess the Efficacy and Safety of Cobitolimod as an add-on to Current Practice in Chronic Active Treatment Refractory Ulcerative Colitis Patients
Brief Title: The Efficacy and Safety of Cobitolimod (Kappaproct®) in Chronic Active Treatment Refractory Ulcerative Colitis Patients
Acronym: COLLECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InDex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSUC-01/10; 2011-003130-14 (EudraCT Number)
Record Dates: First submitted 2011-12-12; First posted 2011-12-16 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Colitis, Ulcerative
Keywords: Colitis, Ulcerative; Gastrointestinal Diseases; Inflammatory Bowel Diseases; Immunomodulatory Therapy; Glucocorticoids; Anti-Inflammatory Agents; Therapeutic uses
MeSH Terms: conditions — Colitis, Ulcerative; Gastrointestinal Diseases; Inflammatory Bowel Diseases | interventions — cobitolimod; DIMS0150

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cobitolimod (Experimental): 2 doses 4 weeks apart
  Interventions: Drug: Cobitolimod
- Placebo (Placebo Comparator): 2 doses 4 weeks apart
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cobitolimod — 30 mg rectal dose at week 0 and 4
  Other Names: DIMS0150, Kappaproct
  Arms: Cobitolimod
Drug: Placebo — Rectal dose at week 0 and 4
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if cobitolimod (former called Kappaproct®) is effective in the treatment of chronic active ulcerative colitis patients not responding to available therapy.

DETAILED DESCRIPTION:
The study is a placebo-controlled, double-blind, randomised study to assess the efficacy and safety of cobitolimod as an add-on to current practice in treatment refractory ulcerative colitis patients. The study population will be chronic active ulcerative colitis patients who are no longer responding adequately to standard therapies and who are potential candidates for colectomy. Cobitolimod/placebo will be add-on treatment allowing all included patients to be on concomitant medication, as well as mandatory steroids at inclusion, throughout the study.

Cobitolimod (DIMS0150) is a modified single strand DNA-based synthetic oligodeoxyribonucleotide of 19 bases in length. The drug functions as an immunomodulatory agent by targeting the Toll-like receptor 9 (TLR9) present in immune cells (i.e., B-cells and pDCs) residing in high abundance on mucosal surfaces, such as colonic and nasal mucosa. The mucosa of the colon and rectum of patients with ulcerative colitis contains active immune cells, which produce damage to the tissue. The activation of these cells by cobitolimod results in the systemic release of specific cytokines (e.g., IL-10 and type I interferons) and chemokines which are believed to be important factors for the clinical effect cobitolimod of cobitolimod. 131 eligible patients was randomly assigned in a 2:1 allocation to receive two single rectal doses of cobitolimod at 30 mg each, or placebo, at week 0 and 4.

The primary endpoint is the induction of clinical remission at week 12 and patients will be continuously followed for efficacy and safety until 12 months after the first dose. Secondary endpoints include the induction of symptomatic remission (number of stools and blood in stools), induction of registration remission (clinical and endoscopic remission) and rate of colectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Well established diagnosis of moderate to moderately severe chronic active UC with a CAI score ≥9, an endoscopic score ≥2, not responding adequately to currently available therapies and potential candidates for colectomy. Previously tried therapies should include:

   * At least one treatment course with mesalazine; at least 2.4 g/day for at least 4 weeks, or at least one treatment course with similar drugs in this class.
   * At least one full dose treatment course of corticosteroids (which can be the treatment of a recent relapse), with up to 0.75 mg/kg as a starting dose or highest dose according to local clinical practice.
   * At least one treatment course of azathioprine or mercaptopurine of at least 3 months duration and/or at least one adequate treatment course of an anti-TNF alpha.
   * Any unsuccessful combination treatment of the above.
   * May have tried treatment with cyclosporine and/or tacrolimus or any other immunosuppressant/immunomodulating agent.
   * Intolerance to any of the above medications is judged as inadequate response.
3. Patients shall at study enrolment be on an accumulated stable tolerable GCS dose equivalent to at least 140 mg of prednisolone/prednisone (by any route of administration) for the last two weeks. Patients may also be on concomitant therapies such as, but not restricted to, 5-ASA, azathioprine and sulphasalazine.
4. Ability to understand the treatment, willingness to comply with all study requirements, and ability to provide informed consent.

Exclusion Criteria:

1. Patients with suspicion of Crohn's enterocolitis, ischaemic colitis, radiation colitis, diverticular disease associated colitis, as well as microscopic colitis should be excluded. Patients with disease limited to the rectum (ulcerative proctitis) should also be excluded.
2. History or presence of a clinically significant cardiovascular, hepatic, renal, haematological, endocrine, neurological, psychiatric disease, or immune compromised state as judged relevant by the investigator.
3. Patients with acute fulminant UC and/or signs of systemic toxicity to an extent that requires immediate surgical action.
4. History or presence of any colonic malignancy and/or dysplasia.
5. Concomitant treatment with cyclosporine, tacrolimus, anti-TNFs or similar immunosuppressants/immunomodulators is not allowed and should have been discontinued 4 weeks before enrolment. Patients who fail the wash-out criteria can undergo wash-out and be re-screened at a later time point. Ongoing treatment of anti-TNFs, tacrolimus or similar immunomodulators/immunosuppressant drugs should only be stopped in case of documented lack of efficacy or in case of intolerable side effects.
6. Treatment with antibiotics or Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) within two weeks before enrolment.
7. An active ongoing infection.
8. History of latent or active tuberculosis, evidence of prior or currently active tuberculosis by chest x-ray, patient with or having had frequent close contact with person with active tuberculosis, patients who previously have tested positive for a tuberculin skin test, or Mantoux (PPD) test, except in the case of previous vaccination or positive interferon gamma release test during screening or within 12 weeks prior to randomisation.
9. Known history of HIV infection based on documented history with positive serology or HIV positive serology.
10. Previously documented positive hepatitis B surface antigen determination, determination of total antibodies to the hepatitis B capsid antigen and/or hepatitis C antibody (HCVAb) with confirmation using the ribonucleic acid of hepatitis B virus.
11. Positive Clostridium difficile stool assay.
12. Currently receiving parenteral nutrition or blood transfusions.
13. Pregnancy or breast-feeding.
14. Women of childbearing potential not using reliable contraceptive methods (reliable methods are barrier protection, hormonal contraception, intra-uterine device or abstinence) throughout the duration of the study (52 weeks).
15. Concurrent participation in another clinical study with investigational therapy or previous use of investigational therapy within 30 days before enrolment. Patients who fail the wash-out criteria can undergo wash-out and be re-screened at a later time point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hawkey, MD, Principal Investigator — Nottingham Digestive Diseases Centre, Queens Campus University Hospitals, Nottingham, UK
Locations (37):
- Czechia (7):
  - Site 402, Hradec Králové
  - Site 404, Hradec Králové
  - Site 406, Ostrava
  - Site 407, Ostrava
  - Site 405, Prague
  - Site 409, Prague
  - Site 403, Slaný
- Site 702, Pierre-Bénite, France
- Germany (11):
  - Site 501, Berlin
  - Site 508, Bottrop
  - Site 514, Erlangen
  - Site 510, Frankfurt
  - Site 509, Freiburg im Breisgau
  - Site 504, Hanover
  - Site 511, Herne
  - Site 503, Jena
  - Site 507, Regensburg
  - Site 502, Stade
  - Site 513, Stuttgart
- Hungary (5):
  - Site 205, Békéscsaba
  - Site 204, Budapest
  - Site 207, Budapest
  - Site 203, Kaposvár
  - Site 202, Szekszárd
- Italy (2):
  - Site 302, Rome
  - Site 304, Rome
- Poland (7):
  - Site 604, Krakow
  - Site 605, Lodz
  - Site 607, Lodz
  - Site 606, Rzeszów
  - Site 601, Warsaw
  - Site 602, Warsaw
  - Site 603, Warsaw
- United Kingdom (4):
  - Site 104, Edinburgh
  - Site 102, London
  - Site 103, Norwich
  - Site 101, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atreya R, Reinisch W, Peyrin-Biroulet L, Scaldaferri F, Admyre C, Knittel T, Kowalski J, Neurath MF, Hawkey C. Clinical efficacy of the Toll-like receptor 9 agonist cobitolimod using patient-reported-outcomes defined clinical endpoints in patients with ulcerative colitis. Dig Liver Dis. 2018 Oct;50(10):1019-1029. doi: 10.1016/j.dld.2018.06.010. Epub 2018 Jun 22. PMID 30120066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 162 subjects screened. Whereof 31 did not meet the criteria
Pre-assignment Details: There were131 patients randomly assigned in a 2:1 allocation to receive 2 rectal doses of cobitolimod at 30 mg, or placebo, respectively.
Period: Overall Study
Arm/Group | Cobitolimod | Placebo
Started | 87 | 44
Received Study Drug | 87 | 43
Completed | 55 | 26
Not Completed | 32 | 18
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 15 | 9
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 10 | 4
Not completed — Non-specified | 4 | 4

BASELINE CHARACTERISTICS:
Population: FAS
Groups:
- Total: Total of all reporting groups
Arm/Group | Cobitolimod | Placebo | Total
Number analyzed (Participants) | 81 | 43 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 40 | 116
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (13.88) | 43.1 (12.31) | 41.8 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 11 | 44
  Male | 48 | 32 | 80
Region of Enrollment [Number; unit: participants]
  Czech Republic | 13 | 6 | 19
  Hungary | 13 | 6 | 19
  Poland | 25 | 14 | 39
  Italy | 2 | 3 | 5
  United Kingdom | 8 | 3 | 11
  Germany | 20 | 11 | 31
Summary of CAI score at baseline by treatment group [Mean (Standard Deviation); unit: units on a scale] — Clinical Activity Index (CAI) which consists of a 7 item scale CAi score is a summary score ranging from 0-29 The summary score indicates increasing values with worsening symptoms
  units on a scale | 11.1 (2.2) | 10.8 (2.1) | 11.0 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Induction of Clinical Remission
Description: The induction of clinical remission at week 12, defined as a CAI score of ≤4.(Full Analysis Set)
Time Frame: Week 12
Population: The FAS consited of all randomized patients who met the inclusion criteria (as assessed by the investigator on the inclusion/exclusion criteria form), and received at least 1 dose of study drug (active or placebo), and who had at least 1 post randomization eligible value of the primary efficacy endpoint
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cobitolimod | Placebo
Number analyzed (Participants) | 81 | 43
Percentage of participants | 44.4 [34.1 to 55.3] | 46.5 [32.5 to 61.1]

2. Secondary Outcome: The Time to Colectomy
Description: Median time to colectomy after 1st dose.
Time Frame: Within 12 months
Population: FAS
Measure: Median (95% Confidence Interval); unit: Time
Arm/Group | Cobitolimod | Placebo
Number analyzed (Participants) | 81 | 43
Time | NA [NA to NA] — Median was not reached due to few events | NA [NA to NA] — Median was not reached due to few events

3. Secondary Outcome: The Rate of Colectomy
Description: Percentage of participants undergoing colectomy at 12 months after 1st dose.
Time Frame: at 12 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Cobitolimod | Placebo
Number analyzed (Participants) | 81 | 43
Percentage of Subjects | 4.9 [1.9 to 12.0] | 11.6 [5.1 to 24.5]

4. Secondary Outcome: Steroid Free Remission at 12 Months
Description: Percentage of participants with steroid free remission at 12 months after 1st dose.
Time Frame: at 12 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Cobitolimod | Placebo
Number analyzed (Participants) | 81 | 43
Percentage of Subjects | 32.1 [22.9 to 42.9] | 30.2 [18.6 to 45.1]

5. Secondary Outcome: The Induction of Mucosal Healing
Description: Percentage of participants with induction of mucosal healing, defined as an endoscopic score of 0 or 1, at week 4 and 12.
Time Frame: Week 4 and 12
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Cobitolimod | Placebo
Number analyzed (Participants) | 81 | 43
Percentage of Subjects
  Week 4 | 34.6 [25.1 to 45.4] | 18.6 [9.7 to 32.6]
  Week 12 | 42.0 [31.8 to 52.8] | 41.9 [28.4 to 56.7]

6. Secondary Outcome: The Induction of Symptomatic Remission
Description: Percentage of participants with induction of symptomatic remission, defined as subscores of blood in stool and number of stools weekly not exceeding 0 and 0 or 1, respectively, at week 4 and 12.
Time Frame: Week 4, 12
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Cobitolimod | Placebo
Number analyzed (Participants) | 81 | 43
Percentage of Subjects
  Week 4 | 32.1 [22.9 to 42.9] | 14.0 [6.6 to 27.3]
  Week 12 | 43.2 [33.0 to 54.1] | 32.6 [20.5 to 47.5]

7. Secondary Outcome: The Induction of Registration Remission
Description: Percentage of participants with induction of registration remission, defined as a CAI score of ≤4 and an endoscopic score of 0 or 1, at week 4 and 12.
Time Frame: Week 4 and 12
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Cobitolimod | Placebo
Number analyzed (Participants) | 81 | 43
Percentage of Subjects
  Week 4 | 21.0 [13.5 to 31.1] | 4.7 [1.3 to 15.5]
  Week 12 | 30.9 [21.9 to 41.6] | 30.2 [18.6 to 45.1]

ADVERSE EVENTS:
Time Frame: 1 year, 2 weeks
Description: All patients who entered into the study and were treated with at least 1 dose of study drug are included in the safety analysis set.
Arm/Group | Cobitolimod | Placebo
Serious Adverse Events (participants affected / at risk) | 10/87 | 8/43
Other Adverse Events (participants affected / at risk) | 31/87 | 6/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cobitolimod (N=87) | Placebo (N=43)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Acute Coronary syndrome (Cardiac disorders) | 1 | 0
Myocardial Ischemia (Cardiac disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Retinal Veon Thrombosis (Eye disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Perirectal abscess (Gastrointestinal disorders) | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1
Clostridial infection (Reproductive system and breast disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal compression fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Sensory Distrurbance (Nervous system disorders) | 0 | 1
Movement disorder (Nervous system disorders) | 0 | 1
Benign Dysplaisa (Reproductive system and breast disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Epistaxis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cobitolimod (N=87) | Placebo (N=43)
Anemia (Blood and lymphatic system disorders) | 4 | 1
Cushingoid (Endocrine disorders) | 4 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Nasopharyngitis (Infections and infestations) | 5 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Headache (Nervous system disorders) | 5 | 2
Depression (Psychiatric disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No